CLINICAL TRIAL: NCT05149339
Title: Effect of Vitamin D Status on A Disintegrin-like And Metalloprotease With Thrombospondin Type 1 Motif 13 (ADAMTS13) and Interleukin 6 (IL-6) in Patients With Acute Myeloid Leukemia
Brief Title: Vitamin D Effect on A Disintegrin-like And Metalloprotease Thrombospondin1 Motif 13& Interleukin 6 in Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Ashraf Abdelhady, Principal Investigator, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB #5208/13-2-2019
Record Dates: First submitted 2021-11-20; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Acute Myeloid Leukemia; Vitamin D Deficiency; ADAMTS13; Interleukin 6
Keywords: ADAMTS13; Interleukin 6; Vitamin D; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Case subgroup with deficient Vitamin D (No Intervention): Group with deficient Vitamin D < 20 ng/mL No treatment for the Vitamin D deficiency
- Case subgroup with deficient Vitamin D + Vitamin D supplementation (Experimental): Group with deficient Vitamin D + Daily oral dose of Cholecalciferol for 28 days for correcting the deficiency
  Interventions: Drug: Cholecalciferol 2800 I.U. ml oral drops
- Case subgroup with normal Vitamin D (No Intervention): Group with normal Vitamin D level > 20 ng/mL

INTERVENTIONS:
Drug: Cholecalciferol 2800 I.U. ml oral drops — (Cholecalciferol 2800 I.U. ml) Oral Drops 15 ml. supplied with a dropper.
  * Composition:
  Each 1 ml (= 28 drops) of oral solution contains: Vitamin D3 (Cholecalciferol) 2800 I.U., (each drop contains 100 IU of vitamin D3).
  Arms: Case subgroup with deficient Vitamin D + Vitamin D supplementation

SUMMARY:
A Disintegrin-like And Metalloprotease with Thrombospondin type 1 motif 13 (ADAMTS13) deficiency was incriminated in poor prognosis, high probability of serious complications and mortality in acute myeloid leukemia (AML) patients. Interleukin 6 (IL-6) produced from AML blasts decreases Cluster of differentiation 34 positive(CD34+) cells differentiation, and inhibits the ADAMTS13 actions. Vitamin D "as an Immune-modulator" inhibits the pro-inflammatory cytokines including IL-6. So, supplementation of vitamin D might help down regulation of interleukin-6 production.

Aim of the study To evaluate the potential relation between Vitamin D status, ADAMTS13 and IL-6 in AML patients.

Objectives

1. Assess Vitamin D level in AML patients
2. Assess ADAMTS13 and IL-6 in AML patients
3. Correlate between Vitamin D level and both of ADAMTS13 and IL-6

DETAILED DESCRIPTION:
I. Setting The study will be carried out in wards of ZAGAZIG University Hospitals II. Subjects The study will be conducted on patients with de novo diagnosis with acute myeloid leukemia III. Inclusion criteria

1. Patient's consent to share in the study
2. Patients' age >18 years
3. Patients with de novo acute myeloid leukemia IV. Exclusion criteria

1. Patients refusing to share in the study 2. Non-Egyptian patients 3. Patients' age < 18 years 4. Pregnant women 5. Patient's with other malignancies 6. Patients with known congenital thrombotic/ hemorrhagic diseases 7. Patients with Thrombotic Thrombocytopenic Purpura 8. Patients with auto-immune diseases

V. Study Design This is a Non-randomized control trial I. Sample size up Finding that ADAMTS13 level in AML patients before treatment is 455+_120 ng/ml versus 570+_100 ng/ml after treatment, the sample was calculated to be 30 patients, 15 patients in each group by using (open EPI) at confidence level 95 and power 80 I. Activities Patients attending to ZAGAZIG University Hospitals. Upon agreement, every patient will be asked to provide written informed consent according to the Declaration of Helsinki of 1979.

All patients will be subjected to the following:

1. Full History taking through an interview
2. Clinical examination
3. Laboratory investigations including:

   1. Complete blood picture ( CBC) using ( Sysmex XS 500)
   2. Peripheral blood film examination
   3. Erythrocyte sedimentation rate ( Westergren tubes )
   4. Prothrombin time, Partial thromboplastin time (Sysmex CS)
   5. C-reactive protein , Liver function tests & Kidney function tests (Roche Diagnostics, Cobas 8000 c702, Switzerland)
   6. Hepatitis C virus antibody, Hepatitis B virus surface antigen and Human deficiency virus antibody
   7. Diagnosis of Acute myeloid leukemia according to clinical findings, CBC, peripheral blood film examination, Bone marrow aspiration, Immunophenotyping (a FACSCAN, Becton Dickinson, San Jose, California, USA)and Cytogenetic analysis.
4. Measuring IL-6 and ADAMTS13 using (Luminex Corporation, Luminex® 200 trademark , Austin, USA) before and after induction therapy
5. Measuring Vitamin D serum level using (Roche Diagnostics, Cobas 6000 e 601, Switzerland) before and after induction therapy and vitamin D supplementation based on its deficiency.
6. Radiology:

   * Echocardiogram
   * Abdominal ultrasound ( If needed)
   * Chest X-Ray II. Data collection Demographic data of the patients will be recorded including name, age, sex and residence. In addition, careful history taking and clinical examination will be done, and data will be registered in special form III. Statistical analysis Our study will be carried on 30 patients with de novo AML. Subjects will be divided into (2) groups as regard treatment of Vitamin D deficiency at the onset of AML diagnosis. Vitamin D therapy will be given to 15 deficient subjects for one month with the recommended doses. All the analytes will be assayed before and after the induction chemotherapy course. Both of these groups will be compared statistically using Statistics program smart solution 22 (SPSS22).

Administrative design:

Approval will be asked from ZAGAZIG University Institutional Review Board (IRB).

C. Ethical considerations

1. The study group will be informed about the nature and the purpose of the study and informed consent will be taken.
2. The study group will not be exposed to any harm or risk.
3. Patient's data will be confidential.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's consent to share in the study
2. Patients' age >18 years
3. Patients with denovo acute myeloid leukemia

Exclusion Criteria:

1. Patients refusing to share in the study
2. Non-Egyptian patients
3. Patients' age < 18 years
4. Pregnant women
5. Patient's with other malignancies
6. Patients with known congenital thrombotic/ hemorrhagic diseases
7. Patients with Thrombotic Thrombocytopenic Purpura
8. Patients with auto-immune diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
(Cholecalciferol 2800 I.U. /ml) Oral drops for Vitamin D deficiency correction | Oral daily dose for 28 days
  Using 1ml of Cholecalciferol as daily Oral drops for 28 days to correct the Vitamin D deficiency in acute myeloid leukemia patients.
  On day 1;The patient is considered deficient with serum Vitamin D level measuring < 20ng/ml using serum samples operated on (Roche Diagnostics, Cobas 6000 e 601, Switzerland) On using the drug for 28 days and measuring the Vitamin D level on the day 28, Vitamin D is considered to be "corrected" with levels > 20 ng/ml

OTHER OUTCOMES:
Serum Vitamin D status effect on ADAMTS13 level in AML patients | 28 days
  Serum Vitamin D (ng/ml) measured using (Roche Diagnostics, Cobas 6000 e 601, Switzerland) on day 1 and day 28 . ADAMTS13 (ng/ml) is measured using (Luminex Corporation, Luminex® 200TM , Austin, USA) on day 1 and day 28 The inter-relation ship will be statistically assessed
Serum Vitamin D status effect on IL-6 level in AML patients | 28 days
  Serum Vitamin D (ng/ml) measured using (Roche Diagnostics, Cobas 6000 e 601, Switzerland) on day 1 and day 28 . IL-6 (PG/ml) is measured using (Luminex Corporation, Luminex® 200TM , Austin, USA) on day 1 and day 28 The inter-relation ship will be statistically assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Dina Ashraf Abdelhady, Cairo, Madinaty, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Liu C, Zhao L, Zhao J, Xu Q, Song Y, Wang H. Reduced ADAMTS-13 level negatively correlates with inflammation factors in plasma of acute myeloid leukemia patients. Leuk Res. 2017 Feb;53:57-64. doi: 10.1016/j.leukres.2016.12.004. Epub 2016 Dec 20. PMID 28033504
- [Result] Liu C, Han M, Zhao L, Zhu M, Xu Q, Song Y, Wang H. ADAMTS-13 activity reduction in plasma of acute myeloid leukemia predicts poor prognosis after bone marrow transplantation. Hematology. 2019 Dec;24(1):129-133. doi: 10.1080/10245332.2018.1532648. Epub 2018 Oct 16. PMID 30322352
- [Result] Cohen-Hagai K, Rashid G, Einbinder Y, Ohana M, Benchetrit S, Zitman-Gal T. Effect of Vitamin D Status on Von Willebrand Factor and ADAMTS13 in Diabetic Patients on Chronic Hemodialysis. Ann Lab Med. 2017 Mar;37(2):155-158. doi: 10.3343/alm.2017.37.2.155. PMID 28029003
- [Result] Zhang Y, Leung DY, Richers BN, Liu Y, Remigio LK, Riches DW, Goleva E. Vitamin D inhibits monocyte/macrophage proinflammatory cytokine production by targeting MAPK phosphatase-1. J Immunol. 2012 Mar 1;188(5):2127-35. doi: 10.4049/jimmunol.1102412. Epub 2012 Feb 1. PMID 22301548
- [Result] Sun X, Cao ZB, Zhang Y, Ishimi Y, Tabata I, Higuchi M. Association between serum 25-hydroxyvitamin D and inflammatory cytokines in healthy adults. Nutrients. 2014 Jan 2;6(1):221-30. doi: 10.3390/nu6010221. PMID 24451309
- [Result] Sun CF, Zhao X, Han F, Jia Q, Wang L, Lu G, Ding HF. [Changes of ADAMTS13 Activity and TSP1 Level in Patients with Hematologic Malignancies]. Zhongguo Shi Yan Xue Ye Xue Za Zhi. 2016 Oct;24(5):1294-1298. doi: 10.7534/j.issn.1009-2137.2016.05.002. Chinese. PMID 27784345
- [Derived] Abdelhady DA, Azab MMM, Alnagar AA, Said N. Effect of vitamin D status on a disintegrin-like and metalloprotease with thrombospondin type 1 motif 13 (ADAMTS13) and interleukin 6 in patients with acute myeloid leukaemia. Eur J Med Res. 2025 Jul 16;30(1):637. doi: 10.1186/s40001-025-02879-8. PMID 40671161